CLINICAL TRIAL: NCT00307463
Title: Effects of Strict Volume Control in Hypertensive Hemodialysis Patients on Cardiac Structure and Chronic Inflammation: a Randomised, Prospective and Controlled Study
Brief Title: Effects of Strict Volume Control in Hypertensive Hemodialysis Patients on Cardiac Structure and Chronic Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ercan OK, professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ege1336
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: End-stage Renal Disease
Keywords: end-stage renal disease; hemodialysis; volume control; ultrafiltration; inflammation; cardiovascular disease; left ventricular hypertrophy; dietary salt restriction
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation; Cardiovascular Diseases; Hypertrophy, Left Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- strict volume control policy (Active Comparator): strict volume control policy: Antihypertensive medicine will be stopped and strict volume control policy will be applied.
  Interventions: Procedure: strict volume control policy
- antihypertensive drugs administration (Other): antihypertensive drugs administration: Antihypertensive medicine will be continued. Target BP will be 130/80 mmHg in both groups.
  Interventions: Procedure: antihypertensive drugs administration

INTERVENTIONS:
Procedure: strict volume control policy — strict volume control by UF and dietary salt restriction
  Arms: strict volume control policy
Procedure: antihypertensive drugs administration — continue antihypertensive medications
  Arms: antihypertensive drugs administration

SUMMARY:
This study aims mainly to investigate the effects of two approaches to control blood pressure in hypertensive hemodialysis patients; using antihypertensive drugs versus strict volume control (by strict dietary salt restriction and persistent ultrafiltration) without using antihypertensive drugs on cardiac structure and inflammation.

DETAILED DESCRIPTION:
This randomised, controlled and prospective study aims mainly to investigate the effects of two approaches to control blood pressure in hypertensive hemodialysis patients; using antihypertensive drugs versus persistent strict volume control without using antihypertensive drugs on cardiac structure (mainly left ventricular hypertrophy)and inflammation.

We hypothesize that better blood pressure control and regression of left ventricular mass may be reached by a policy of strict volume control consisting of strict dietary salt restriction and persistent ultrafiltration.

258 Hypertensive hemodialysis patients (BP>130/80 mmHg and/or being on antihypertensive medication) will be randomized to two arms:

Group 1: Antihypertensive medicine will be stopped and strict volume control policy will be applied.

Group 2: Antihypertensive medicine will be continued. Target BP will be 130/80 mmHg in both groups.

The patients will be evaluated at 12 months for primary outcomes. Primary end-points are significant changes in left ventricular hypertrophy and left ventricular mass and significant change in left ventricular end-diastolic volume.

Secondary end-points are changes in post-dialysis weight, changes in hematocrit, albumin, BNP and hsCRP levels.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-70 years old
* on maintenance bicarbonate hemodialysis scheduled thrice weekly, at least 12 hours/week
* willingness to participate in the study with a written informed consent.

Exclusion Criteria:

* to be scheduled for living donor renal transplantation
* to have serious life-limiting co-morbid situations; namely active malignancy, active infection, end-stage cardiac, pulmonary, or hepatic disease; pregnancy or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2005-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
regression of left ventricular hypertrophy | one year
regression of left ventricular mass | one year
change in left ventricular end-diastolic volume | one year

SECONDARY OUTCOMES:
change in post-dialysis weight, changes in hematocrit, albumin, changes in BNP and hsCRP levels | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Ok, M.D, Study Chair — Ege University School of Medicine Nephrology Department
Locations (2):
- Turkey (Türkiye) (2):
  - Adana Numune Research and Education Hospital, Adana, Adana
  - Ege University School of Medicine Division of Nephrology, Bornova, İzmir